CLINICAL TRIAL: NCT01586637
Title: Assessment of Art Therapy Program for Women With Fibromyalgia: Randomized, Controlled, Blinded Study
Brief Title: Art Therapy to Treat Women With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Andréia S Baptista, PT, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0206/10
Record Dates: First submitted 2012-02-16; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Art Therapy; Pain; Quality of life; Body Image
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Art Therapy; Rehabilitation; Exercise; Physical Therapy Modalities; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Art Therapy (Experimental): This group performed dance classes and regarding the art therapy they have art classes where they learn how to use the drawing to express feelings. The classes were twice a week.
  Interventions: Other: Art Therapy
- Walking (Experimental): The group walked twice a week during one hour.
  Interventions: Other: Walking

INTERVENTIONS:
Other: Art Therapy — This group performed dance classes and regarding the art therapy they have art classes where they learn how to use the drawing to express feelings. The classes were twice a week.
  Other Names: Rehabilitation, exercise, physical therapy
  Arms: Art Therapy
Other: Walking — The group walked twice a week during one hour.
  Other Names: Rehabilitation, exercise, physical therapy
  Arms: Walking

SUMMARY:
Effectiveness of an art therapy program for the treatment of pain and improvements in both quality of life and body image of patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic non-inflammatory syndrome characterized by diffuse pain throughout the body, sleep disorder, stiffness, fatigue, depression and other psychological problems. Patients with FM feel incapable of performing the majority of activities of daily living. Medication offers only short-term benefits. Thus, it is necessary to include other measures for treatment, such as physical activity and patient education. Art therapy combine the field of psychology with artistic activities, working with therapeutic and instructive aspects as well as the potential for personal growth contained in all forms of art.

ELIGIBILITY:
Inclusion Criteria:

* Classification of fibromyalgia by ACR criteria (Wolf et al, 1990)
* Females
* Without distinction of race
* Age 18 to 65 years
* Do not have changed treatment for fibromyalgia for at least 3meses
* signing the consent form

Exclusion Criteria:

* Other ostearticulares rheumatic and painful
* Decompensated cardio-respiratory diseases
* Perform physical activity more than 2x a week for more than 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain | baseline, after 10 weeks, 20 weeks and 40 weeks
  Evaluated with the visual analogue scale

SECONDARY OUTCOMES:
Change in fibromyalgia impact | Baseline, after 10, 20 and 40 weeks
  Evaluated using the Fibromyalgia Impact Questionnaire
Change in Quality of life | Baseline, after 10, 20 and 40 weeks
  Evaluated using the SF-36 questionnaire
Change in Body image | Basline, after 10, 20 and 40 weeks
  Evaluated using the Body Dismorphic Disorder Examination (BDDE) questionnaire
Change in Functional capacity | Baseline, after 10, 20 and 40 weeks
  Evaluated using the six minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Andréia S Baptista, PT, MSc, Principal Investigator — Federal University of São Paulo
Locations (1):
- Andréia Salvador Baptista, São Paulo, São Paulo, Brazil